CLINICAL TRIAL: NCT03846947
Title: Novel MRI Sequence MR Fingerprinting in Breast MRI Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LCCC1853
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Results first posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-04

CONDITIONS: Breast Screening

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- All participants (Experimental): All participants will receive the investigational MR Fingerprinting sequence.
  Interventions: Device: MR Fingerprinting

INTERVENTIONS:
Device: MR Fingerprinting — The MR fingerprinting technique requires less than 15 minutes total and will be added before and after the standard MRI sequence.

SUMMARY:
The purpose of this study is to evaluate potential clinical efficacy of a novel magnetic resonance imaging (MRI) approach, MR fingerprinting, capable of providing quantitative measures of important tissue properties, which could provide important insights into normal breast tissue. This new MRI sequence will be added to the screening breast Dynamic Contrast Enhanced (DCE) MRI for high risk normal patients.

DETAILED DESCRIPTION:
This is a feasibility study of the use of the additional MR fingerprinting (MRF) scanning sequence with a total of 12 minutes scanning time to our clinical screening breast DCE MRI examination before contrast medium injection and at the end of scan. This additional scanning sequence may provide faster and better quantitative tissue characterization comparing to conventional MR sequences. There is no investigational contrast agent in this study. We propose that the additional MRF sequence may provide faster and more accurate tissue characteristics imaging for clinical evaluation of breast tissue. Patients will be enrolled in with scheduled high risk screening DCE MRI (n=30). The MR imaging will be performed in the clinical 1.5T MR scanners in UNC as normally done for the patients MRI schedule. We only add an additional MRF sequence within the MRI exam just prior to the contrast enhancement scan.

Quantitative measurement of the breast tissue will be performed after the MR exam. The region-of-interest (ROI) of normal breast parenchyma was recorded. The ROI will be saved and encoded to the T1 map, T2 map in MRF, T1 weighted imaging, T2 weighted imaging. A large variety of imaging ROI-based quantitative measures will be calculated among normal glands in bilateral breasts to evaluate different ROI characteristics among different patients and between bilateral breasts in each patient.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking patients
* Ages 18 to 99 years old
* Scheduled to undergo a screening breast MRI study
* Capable and willing to provide signed informed consent

Exclusion Criteria:

* Claustrophobia
* Presence of pacemaker, intracranial aneurysm clip, bladder stimulator, cochlear implant or metal near eyes or near pelvis that would create excessive imaging artifact
* Known hypersensitivity to contrast agent or to any component of contrast agent refractory to standard medications (antihistamines, steroids)
* Impaired kidney function (serum creatinine level > 1.8 mg/dl or a glomerular filtration rate < 60 as approximated using serum creatinine levels) unless anuric and on dialysis.
* Inability to tolerate MRI (e.g., inability to lie flat for >1 hour)
* Pregnancy or lactating female
* Previous history of mastectomy or lumpectomy
* Breast enhancements (i.e. implants)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cherie Kuzmiak, DO,FACR,FSBI, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 28
Completed | 26
Not Completed | 2
Not completed — technical issues with imaging sequence | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.98 (13.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Intensity Score of Normal Breast Tissue for Left Breast Tissue Compared to Right for T1 Imaging Sequence
Description: The normal breast tissue intensity value from the MRI will be used to compare between sides in same patient in the T1 sequence. The ratio of the left intensity score to the right intensity score will be averaged. The intensity value is a quantitative measurements of T1 relaxation time, an intrinsic magnetic tissue property that is correlated with a variety of pathological conditions.
Time Frame: during MRI, approximately 1 hour
Population: Two participants did not undergo the investigational sequence due to technical errors with the sequence at the time of the scan.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | All Participants
Number analyzed (Participants) | 26
ratio | 1.07 (0.23)

2. Primary Outcome: Ratio of Intensity Score of Normal Breast Tissue for Left Breast Tissue Compared to Right for T2 Imaging Sequence
Description: The normal breast tissue intensity value from the MRI will be used to compare between sides in same patient in the T2 sequence. The ratio of the left intensity score to the right intensity score will be averaged. The intensity value is a quantitative measurements of T2 relaxation time, an intrinsic magnetic tissue property that is correlated with a variety of pathological conditions.
Time Frame: during MRI, approximately 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | All Participants
Number analyzed (Participants) | 26
ratio | 1.03 (0.24)

3. Primary Outcome: Ratio of Intensity Score of Normal Breast Tissue for Left Breast Tissue Compared to Right for the Investigational (MRF) Imaging Sequence
Description: The normal breast tissue intensity value from the MRI will be used to compare between sides in same patient in the investigational (MRF) sequence. The ratio of the left intensity score to the right intensity score will be averaged. The intensity value is a quantitative measurements of MRF relaxation time.
Time Frame: during MRI, approximately 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | All Participants
Number analyzed (Participants) | 26
ratio | 1.08 (0.17)

ADVERSE EVENTS:
Time Frame: 30 minutes post imaging, up to 1 hour
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT03846947/Prot_SAP_000.pdf